CLINICAL TRIAL: NCT00600314
Title: Measurements of Resting Energy Expenditure in Patients With or at Risk of Developing Graft Versus Host Disease
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: SCT 0405 REE
Record Dates: First submitted 2008-01-08; First posted 2008-01-24 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Graft-Versus-Host Disease
Keywords: Graft-Versus-Host Disease; Transplantation, Allogeneic; Transplantation, Hematopoietic Stem Cell; Calorimetry, Respiration
MeSH Terms: conditions — Graft vs Host Disease; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High risk: Patients who are at high risk of developing acute or chronic GVHD
- GVHD: Patients who currently have either grade II or greater acute GVHD, or clinically extensive chronic GVHD

SUMMARY:
This study aims to show that the MedGem indirect calorimetry measurement device will be feasible to use in children with GVHD. Also, it aims to show that children with chronic GVHD will have elevated REE that is not adequately predicted by standard equations.

DETAILED DESCRIPTION:
Chronic Graft versus Host Disease (GVHD) is an important cause of morbidity and mortality in patients undergoing allogeneic bone marrow and hematopoietic progenitor cell transplantation. In adults, it has been shown that patients with acute or chronic GVHD have an increase in their resting energy expenditure (REE), likely as a result of chronic systemic inflammation. These studies have not yet been performed in children. This study's objective is to determine the REE of pediatric patients with acute and chronic GVHD after hematopoietic stem cell transplantation (HSCT).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 7-30 years of age
* Signed informed consent
* One of the following three criteria must be met:

  * Presence of grade II or greater acute GVHD as defined by Keystone criteria
  * Presence of clinically extensive chronic GVHD as defined by the revised Seattle criteria
  * Any subject identified prior to allogeneic transplant, or following allogeneic transplant, who is at risk for acute or chronic GVHD

Exclusion Criteria:

* Inability to meet the requirements of the study procedures
* Any subject who is receiving supplemental oxygen
* Withdrawal of consent

Ages: 7 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: High risk population: patients who are at high risk of developing acute or chronic Graft versus Host Disease (GVHD) following an allogeneic transplant.
  GVHD population: patients with active GHVD, either acute or chronic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Feasibility - can the procedure be adequately performed in a child? | Spring of 2010

SECONDARY OUTCOMES:
Measure of resting energy expenditure - kcal/day and oxygen consumption (VO2 mL/min) | Spring of 2012

CONTACTS AND LOCATIONS:
Overall Officials: Morris Kletzel, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States